CLINICAL TRIAL: NCT05738005
Title: DRITA Pilot Trial: Dietary Reporting in the Amyloidoses
Brief Title: Dietary Reporting in the Amyloidoses
Acronym: DRITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Multiple Myeloma Multidisciplinary team leader, M.D., Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-067
Record Dates: First submitted 2023-01-20; First posted 2023-02-21 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tracking Dietary/Supplement Intake on MyFitnessPal smartphone application (app) (Other): MyFitnessPal smartphone application is used to track daily dietary intake and herbal/alternative supplements.
  Interventions: Other: Tracking Dietary/Supplement Intake on MyFitnessPal smartphone application (app)

INTERVENTIONS:
Other: Tracking Dietary/Supplement Intake on MyFitnessPal smartphone application (app) — Amyloidosis patients will use MyFitnessPal application to track dietary intake and use of herbal/alternative supplements in from week 2-9. Patient's usage of the application and questionnaires completed by the patient at the start, Week 2 and Week 10 will determine feasibility.

SUMMARY:
The goal of this clinical trial is to learn about malnutrition and weight loss in patients with Amyloidosis.

The main question it aims to answer is:

Is it feasible to use a low-cost nutrition-based application (apps) for use on a smartphone to obtain detailed information on caloric intake in Amyloidosis patients

Participants will be asked to:

* Download the MyFitnessPal application on their smartphone and view an online tutorial
* After a week of practice, from weeks 2-9, participants will enter daily dietary intake as well as daily herbal/alternative supplement intake into the MyFitnessPal application on their smartphone.
* complete a questionnaire prior to starting the application, after week 2 and at week 10 after starting the application

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with any type of amyloidosis
* Speak, read and write in English
* Willing to use the MyFitnessPal app on their own smartphone

Exclusion Criteria:

* a planned autologous stem cell transplant or a solid organ transplant in the 12 weeks after enrollment
* cognitive or perceptual disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Adherence Rate | 56 days
  The adherence is defined by the status (yes vs. no) of data recording per day; The adherence rate will be calculated by the ratio of the number of days of adherence to the total number of days of trial (i.e., 56 days); The status of data recording per day will be considered 'yes' if the participant completes a daily survey.

SECONDARY OUTCOMES:
Subsequent adherence rate | 63 days (= 56 days + Week 10)
  The subsequent adherence is the status of data recording per day during the third phase (Week 10) of trial participation (i.e., 7 days); The subsequent adherence rate will be calculated by the ratio of the number of days of adherence during the third phase (Week 10) of trial participation (i.e., 7 days); The status of data recording per day will be considered 'yes' if the participant completes a daily survey.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zonder, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No